CLINICAL TRIAL: NCT01619436
Title: The Effect of Clonidine in Glycemia During Coronary Artery Bypass Graft With Cardiopulmonary By-pass.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Marcello F Salgado Filho, MD, Principal investigator, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0279/03.05.2010
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Glycemia During Coronary Artery Bypass Graft; Sedation During Pre-anesthetic Medication
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clonidine (Active Comparator): clonidine 2 mg/kg IV
  Interventions: Drug: Clonidine
- ringer lactato 1 ml (Placebo Comparator): Ringer lactato 1 ml IV as Placebo
  Interventions: Drug: Ringer lactato

INTERVENTIONS:
Drug: Clonidine — bolus, clonidine 2 mg/kg IV
  Arms: clonidine
Drug: Ringer lactato — 1 ML ringer lactato IV, as placebo
  Arms: ringer lactato 1 ml

SUMMARY:
The purpose of this study is the randomized blind research of the assessment of the different levels of glycemia during Coronary Artery Bypass Graft (CABG) with cardiopulmonary by-pass (CPB) between clonidine and placebo. As clonidine decrease the inflammatory response during cardiac surgery, the investigators would like to know if the glycemia levels in clondine group will be lower than placebo group.

ELIGIBILITY:
Inclusion Criteria:

* elective CABG EF > 40% Sinus ritmy

Exclusion Criteria:

* precordialgia emergency surgery combinated surgery not agreement

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
sedation | 2 years
  Clonidine 2 mg/kg IV. assessment sedation with Ransay scale

SECONDARY OUTCOMES:
Glycemia | 2 years
  clonide 2 mg/kg. assessment the glycemia during CPB.

CONTACTS AND LOCATIONS:
Locations (1):
- National institut of Cardiology, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- See also: Related Info — http://www.sba.com.br
- See also: Related Info — http://www.capes.com.br
- See also: Related Info — http://www.rba.com.br
- See also: Related Info — http://www.ovidsp.com